CLINICAL TRIAL: NCT06583499
Title: Investigating The Effect Of Transtheoretical Model Based Nutrition Education On Sustainable Dietary Behaviour In Adolescents
Brief Title: Effect of Transtheoretical Model Based Nutrition Education on Sustainable Nutrition Behavior in Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ozlem Muslu, research scientist, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ErciyesU-DYT-OM-01
Record Dates: First submitted 2024-05-05; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Nutrition, Healthy
Keywords: Healthy Nutrition; Education; Diet, Food, And Nutrition; Transtheoretical Model; Transtheoretical Model Of Behavior Change; Adolescent Nutrition Sciences

STUDY DESIGN:
Intervention Model Description: There are two groups: the study group, which will receive educational intervention, and the control group, which will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (educated about sustainable nutrition) (Experimental): The research will be conducted in an Anatolian high school. The experimental group will be randomly selected from the students who meet the inclusion criteria and are willing to participate in the study. The experimental group will receive sustainable nutrition education programme based on the transtheoretical model. The training content will be applied face-to-face at most twice a week for five weeks.
  Interventions: Behavioral: Sustainable nutrition education based on the transtheoretical model
- Control Group ( non-educated about sustainable nutrition) (No Intervention): In order to prevent any potential influence from peer interaction, the control group will be composed of students from another Anatolian high school with a similar socio-economic and educational background. The control group will be randomly selected from students who meet the inclusion criteria and are willing to participate in the study. The sustainable nutrition education programme will not be applied to this group.

INTERVENTIONS:
Behavioral: Sustainable nutrition education based on the transtheoretical model — Before the intervention begins, the Sustainable Nutrition Behaviour Change Stage Survey will be administered to determine participants' training stage. In addition, the Transtheoretical Model (TTM) Based Sustainable Nutrition Scales will be administered to evaluate the effectiveness of the training programme.
  TTM Based Nutrition Training Programme consists of 11 modules developed according to the stages of the model.The methodology and tools used are aligned with the objectives of the training programme.The training modules are offered twice a week, with each session lasting a maximum of 40 minutes and continues for a total of 5 weeks. Participants may attend more than one training session in order to develop behaviours that increase adherence to a sustainable diet. At the end of the training programme, data from the Transtheoretical Model-Based Sustainable Nutrition Behaviour Scale will be collected again and evaluated by comparison with the baseline data set..
  Arms: Intervention Group (educated about sustainable nutrition)

SUMMARY:
The aim of this intervention study is to evaluate the effect of sustainable nutrition education based on the Transtheoretical Model (TTM) on adolescent behavior.

The main questions to be answered are:

* Do adolescents have sufficient knowledge about sustainable nutrition?
* Can a sustainable nutrition education based on TTM lead to positive changes in the sustainable eating habits of adolescents?

Researchers will compare the study group that received the education with the control group that did not receive the education to determine the effect of TTM based nutrition education on dietary behavior.

Participants will:

* Receive education relevant to the behavior change phase.
* Receive a maximum of two training sessions per week, and the training will last 5 weeks.

DETAILED DESCRIPTION:
Sustainable diets are essential for maintaining health and meeting the nutritional needs of future generations. Adolescents, who make up over 16% of the world's population, play a crucial role in achieving the 2030 Sustainable Development Goals. Adolescent health is essential for maintaining maternal and child health, reducing quality of life, and life expectancy. Traditional interventions, such as health education, are less effective than theory-based methods. The transtheoretical model has been reported as a successful strategy for nutrition interventions aimed at improving dietary behavior among adolescents, highlighting the importance of ensuring adolescents have the right eating habits and adequate nutrition for a healthy society.

This study was planned to examine the effect of TTM-based sustainable nutrition education on behaviour in adolescents. Permission was obtained from the Ministry of National Education for the study.

The study group (n = 35), which will receive the educational intervention, will be randomly selected from 9th grade students studying at high school in Ankara who agree to participate in the study. The control group (n = 35), which will not receive educational intervention, will be randomly selected among 9th grade students who are studying at another high school with a similar socioeconomic and educational level and who agree to participate in the study in order to prevent peer interaction.

Before the educational intervention, the researcher will apply the prepared questionnaire form to both the control group and the study group using the face-to-face interview technique. In addition, the Transtheoretical Model of Sustainable Nutrition Behaviour Change Stage Question will be asked, the behavior stage of the participants will be determined, and the Transtheoretical Model of Sustainable Nutrition Behaviour Scales will be applied.

In the second phase of the study, the working group will participate in the Transtheoretical Model-Based Sustainable Nutrition Education Programme. The training will take place twice a week in sessions of 35 to 40 minutes each. The training will last 5 weeks.

In the final phase of the study, the prepared questionnaire form, the Transtheoretical Model Sustainable Nutrition Behaviour Change Stage Questionnaire and the Transtheoretical Model of Sustainable Nutrition Behaviour Scales will be administered to both the control and study groups.

ELIGIBILITY:
Inclusion Criteria:

* Being in the ninth grade
* Read the consent form and mark the phrase "I accept" in the form.
* Being between the ages of 14-18
* Food insecurity raw score is less than 2

Exclusion Criteria:

* Being in the 10th, 11th, 12th grade
* Refusing to participate in the study
* Food insecurity raw score is less than 2
* Being on a special diet due to a health problem

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-12-07 (Estimated)

PRIMARY OUTCOMES:
Change in Transtheoretical Model Based Sustainable Nutrition Behaviour Scales | baseline and week 5
  The scale consists of 44 items. It is a 5-point Likert type scale. Evaluation is made on a scale from 1 to 5, from never to always.As scores increase, behavioral changes towards sustainable and healthy eating, decision-making, and self-efficacy develop in a positive direction.
Change in Transtheoretical Model Based Sustainable Nutrition Behavior Change Stage Question | baseline and week 5
  Participants will be given a definition of sustainable and healthy nutrition, and they will be asked to evaluate their sustainable and healthy nutrition behaviors according to the definition and to mark which stage they are in according to the TTM change stage.
  Stage of behaviour determined according to the options offered in accordance with the definition:
  Pre-contemplation Stage : (☐) I do not currently eat according to the definition and do not plan to change my diet in the next 6 months.
  Contemplation Stage : ( ☐ ) I do not currently eat according to the definition, but plan to change my diet in the next 6 months.
  Preparation Stage : ( ☐ ) I do not currently eat according to the definition, but I plan to eat healthier and consider the environmental impact in the next 30 days.
  Action Stage : ( ☐ ) I have been on a sustainable eating plan for 6 months now. Maintenance Stage : ( ☐ ) I have been on a sustainable eating plan for over 6 months.

SECONDARY OUTCOMES:
Food security survey for individuals aged 12 and over | baseline
  The survey consists of nine questions. It has a 3-point Likert structure. Responses of "a lot" or "sometimes" are coded as affirmative.The sum of the positive answers given to the questions determines the participant's raw score on the scale.
  * Raw score 0-High food security
  * Raw score 1-Marginal food security
  * Raw score 2-5-Low food security
  * Raw score 6-9-Very low food security
  Low food security and very low food security outcomes are referred to as "food insecure
Change in Sustainable and Healthy Eating Behaviors Scale | baseline and week 5
  The scale consists of 34 items. It is a 7-point Likert type scale. Evaluation is made on a scale from 1 to 7, from never to always.
Change in The Food Frequency Questionnaire (FFQ) | baseline and week 5
  It is a food consumption frequency form with 16 nutrients. Participants were required to indicate the frequency of consumption of the specified foods and meals by selecting one of the following options: "every day (5), 5-6 days a week (4), 3-4 days a week (3), 1-2 days a week (2), 1-2 days a month (1) and never (0)".
Body Mass Index (BMI) | baseline and week 5
  In order to calculate the Body Mass Index (BMI), the height and weight of all participants will be measured.
  Height measurement will be made with a portable height meter supported by the wall with light clothes without shoes, with the head upright, looking straight ahead, the line passing through the eyes and ears parallel to the ground, legs straight and closed, arms at the side, shoulders relaxed, heels, hips and shoulders on the Frankfurt plane against the wall.
  Weight measurement will be done with a 100 g sensitive digital scale.
  BMI will be calculated by dividing weight (kg) by the square of height (m), and age and gender-appropriate percentile values will be determined. A value between the 85th and 95th percentile will be classified as overweight, while a value above the 95th percentile will be classified as obese.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem MUSLU, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)